CLINICAL TRIAL: NCT02456402
Title: Randomized Controlled Trial of Drug Coated Balloon Compared to Bare Metal Stent Using FFR-guidance for the Treatment of de Novo Coronary Artery Lesions
Brief Title: Drug Coated Balloon Compared to Bare Metal Stent for de Novo Coronary Artery Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Prof Eun-Seok Shin, MD. PhD., Interventional Cardiologist, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2015-05-18; First posted 2015-05-28 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Stable Angina; Unstable Angina
MeSH Terms: conditions — Angina, Stable; Angina, Unstable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Coated Balloon (Experimental): PCB (SeQuent Please®, paclitaxel-coated balloon catheter, B. Braun, Melsungen, Germany)
  Interventions: Device: Drug Coated Balloon
- Bare Metal Stent (Active Comparator): BMS (Vision®)
  Interventions: Device: Bare Metal Stent

INTERVENTIONS:
Device: Drug Coated Balloon — If post balloon angioplasty FFR is more than 0.80, either DCB treatment or BMS implantation will be carried out based on randomization of 1:1. DCB (SeQuent Please paclitaxel-coated balloon catheter, B. Braun, Melsungen, Germany) will be applied at the predilated lesions. PCB will be delivered rapidly and inflated for 60 seconds with nominal pressure.
  Arms: Drug Coated Balloon
Device: Bare Metal Stent — BMS (Vision®) will be applied at the predilated lesions after angiographic confirmation of the target lesion.
  Arms: Bare Metal Stent

SUMMARY:
This randomized trial will assess the efficacy of Drug Coated Balloon (DCB) compared to Bare Metal Stent (BMS) using Fractional Flow Reserve (FFR) guidance for de novo coronary artery lesions in patients unable to tolerate dual antiplatelet therapy and at high risk of bleeding. Patients will be randomized after balloon angioplasty to receive either DCB or BMS. Endpoints are late luminal loss at 9 months, and major adverse cardiac events including arterial thrombosis at 1, 9 and 12 months.

DETAILED DESCRIPTION:
Although the use of drug-eluting stents (DES) has reduced in-stent restenosis when compared to bare metal stents (BMS) and decreased the incidence of adverse clinical events (1-2), DES therapy is limited by delayed arterial healing, late acquired malapposition and neo-atherosclerosis leading to an increased risk of late stent thrombosis and late restenosis (3-4). Conceptually, a permanent stent inhibits advantageous vascular remodeling and durable polymer provokes excessive inflammation (5). Non-stent based local drug delivery using paclitaxel-coated balloon has emerged as a new clinical treatment alternative by maintaining the anti-proliferative properties of DES (6). There is limited data on the efficacy of Drug Coated Balloon (DCB) treatment for de novo coronary lesions when compared to BMS. To avoid the risk of abrupt closure of target lesion after balloon angioplasty, a reliable predictor of coronary flow is necessary especially in de novo lesions of major coronary arteries. Therefore, using fractional flow reserve (FFR) after angioplasty as a good indicator of immediate functional improvement and reduced restenosis (7), the aim of this study is to assess the efficacy of DCB treatment compared to BMS in patients with de novo coronary artery lesions.

Patients with de novo coronary artery lesions with > 50% stenosis in a single vessel and at high risk of bleeding with the inability to tolerate dual antiplatelet therapy (DAPT) will be included in this trial. Patients will undergo balloon angioplasty and if the FFR post balloon angioplasty is > 0.80, they will be randomized to receive either DCB or BMS. Patients will receive Quantitative Coronary Angiography (QCA) analysis at 9 months follow-up. Endpoints are late luminal loss at 9 months and major adverse events including arterial thrombosis at 1, 9 and 12 months and these endpoints will be compared between DCB and BMS groups.

ELIGIBILITY:
Inclusion Criteria:

* Stable Angina and Unstable angina
* single de novo coronary artery lesions in a single vessel with > 50% diameter stenosis with a reference diameter > 2.75mm
* Patients at high risk of bleeding and whom cannot tolerate dual antiplatelet therapy for > 1 month are inclusion criteria for the study and are listed here:
* Unexplained anemia
* Atrial fibrillation with CHADSVASC > or equal to 1
* Patients awaiting for non cardiac surgery within a year
* History of massive hemorrhage requiring transfusion
* History of upper GI bleeding
* Malignancy
* Poor compliance with medication

Exclusion Criteria:

* STEMI/NSTEMI within the preceding 72 hours
* Multivessel disease, chronic total occlusion, long lesions and left main disease
* heart failure with ejection fraction < 35% and/or cardiogenic shock
* Previous history of or planned coronary artery bypass grafting
* life expectancy of less than 1 year

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Late luminal loss | 9 months

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) (death, myocardial infarction, repeat revascularization, recurrent ischemic symptoms) | Post procedure (up to 1 hour), 1 month, 9 months and 12 months
Arterial thrombosis | Post procedure (up to 1 hour), 1 month, 9 months and 12 months
  Any stent thrombosis - acute, subacute/late stent thrombosis
Fractional Flow Reserve | Post procedure (up to 1 hour) and 9 months
  FFR is the ratio of the pressure measured at the distal portion of the target lesion and the aortic ostium at maximal hyperemia

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Seok Shin, M.D., PhD., Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

REFERENCES:
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Joner M, Finn AV, Farb A, Mont EK, Kolodgie FD, Ladich E, Kutys R, Skorija K, Gold HK, Virmani R. Pathology of drug-eluting stents in humans: delayed healing and late thrombotic risk. J Am Coll Cardiol. 2006 Jul 4;48(1):193-202. doi: 10.1016/j.jacc.2006.03.042. Epub 2006 May 5. PMID 16814667
- [Background] Nakazawa G, Vorpahl M, Finn AV, Narula J, Virmani R. One step forward and two steps back with drug-eluting-stents: from preventing restenosis to causing late thrombosis and nouveau atherosclerosis. JACC Cardiovasc Imaging. 2009 May;2(5):625-8. doi: 10.1016/j.jcmg.2009.01.011. No abstract available. PMID 19442951
- [Background] Unverdorben M, Kleber FX, Heuer H, Figulla HR, Vallbracht C, Leschke M, Cremers B, Hardt S, Buerke M, Ackermann H, Boxberger M, Degenhardt R, Scheller B. Treatment of small coronary arteries with a paclitaxel-coated balloon catheter in the PEPCAD I study: are lesions clinically stable from 12 to 36 months? EuroIntervention. 2013 Sep;9(5):620-8. doi: 10.4244/EIJV9I5A99. PMID 24058078
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Bech GJ, Pijls NH, De Bruyne B, Peels KH, Michels HR, Bonnier HJ, Koolen JJ. Usefulness of fractional flow reserve to predict clinical outcome after balloon angioplasty. Circulation. 1999 Feb 23;99(7):883-8. doi: 10.1161/01.cir.99.7.883. PMID 10027810
- [Derived] Shin ES, Lee JM, Her AY, Chung JH, Eun Lee K, Garg S, Nam CW, Doh JH, Koo BK. Prospective randomized trial of paclitaxel-coated balloon versus bare-metal stent in high bleeding risk patients with de novo coronary artery lesions. Coron Artery Dis. 2019 Sep;30(6):425-431. doi: 10.1097/MCA.0000000000000755. PMID 31009399